CLINICAL TRIAL: NCT05864326
Title: Effect of Heated Saline in Duration of Cervical Ripening in Women Having Labor Induction With Cervical Balloon: a Randomized Controlled Study
Brief Title: Heated Saline in Cervical Balloon for Labor Induction, a RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Begona Martinez de Tejada (Other)
Responsible Party: Sponsor-Investigator, Begona Martinez de Tejada, Professor, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-02120
Record Dates: First submitted 2023-04-02; First posted 2023-05-18 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Cervical Ripening; Induction of Labor; Unfavorable Cervix; Mechanical Method
Keywords: Cervical ripening; Induction of Labor; Unfavorable cervix; Mechanical method

STUDY DESIGN:
Intervention Model Description: Prospective, single-center, randomized, two-arm, controlled trial, including women requiring cervical ripening during the process IOL using Balloon catheter
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Warm group (Experimental): The Balloon Catheter will be filled with heated saline water up to 40° C
  Interventions: Device: Warm group
- Room temperature group (Active Comparator): the Balloon Catheter will be filled with saline water at room temperature.
  Interventions: Device: Room temperature group

INTERVENTIONS:
Device: Warm group — The operator will introduce a 14Fr or 18Fr Balloon catheter through the cervical canal, up above the internal orifice using a long Pean clamp and inflate the internal balloon with 30 to 80ml of Heated saline water (NaCl 0.9%) at 40°C - according to the mechanic resistance with a graduated syringe.
  Arms: Warm group
Device: Room temperature group — The operator will introduce a 14Fr or 18Fr Balloon catheter through the cervical canal, up above the internal orifice using a long Pean clamp and inflate the internal balloon with 30 to 80ml of unheated saline water (NaCl 0.9%) - according to the mechanic resistance with a graduated syringe.
  Arms: Room temperature group

SUMMARY:
This study is a single-center, randomized, two-arm, controlled trial, including women requiring cervical ripening during the process Induction of Labor using Balloon catheter (BC). The primary objective of the study is to determine if the use of heated saline in the BC used for cervical ripening reduces the length of BC duration.

Participants will be allocated to :

* Intervention or warm group: the BC will be filled with heated saline water up to 40° C
* Standard or room temperature group: the BC will be filled with saline water at room temperature.

DETAILED DESCRIPTION:
Background and Rationale:

Induction of Labor (IOL) is one of the most common interventions in obstetrics. IOL is performed due to fetal, maternal or pregnancy complications to reduce the risk of complication. IOL methods will depend of the state of the cervix at the beginning of the procedure. If cervix is considered unfavorable (Bishop score ≤ 5) an initial phase of ripening is usually proposed. There are various methods of cervical ripening, which can be divided into non-pharmacological (e.g., mechanical methods with transcervical Foley catheter or Cook balloon) and pharmacological (e.g., prostaglandins). IOL can be a long-lasting procedure, especially when cervical ripening is necessary.

Two recent, small studies have shown that the use of warm fluid to inflate the balloon catheter (BC) inserted through the cervix reduces the time of cervical ripening, hence potentially reducing the time of IOL. These results are the only data available regarding the use of saline at different temperatures for inflating the balloon in mechanical methods and show promising effects in terms of reduction in the length of the cervical ripening and labor.

The cervix is mainly composed of collagen. Studies show that the use of heat on connective tissue increase the potential elongation of collagen tissue and the denaturation of this protein.

We hypothesize that the use of heat in the cervical ripening can accelerate the denaturation of the collagen and accelerate the softening of the cervix and therefore reduce the duration of cervical ripening and labor.

Objective(s):

The primary objective of the study is to determine if the use of heated saline in the BC used for cervical ripening reduces the length of BC duration, defined as the time from the insertion to the expulsion or artificial removal of the BC.

The secondary objectives are to evaluate if the use of heated saline compared with room temperature:

1. Decreases the length from the start of the induction until the achievement of a favorable cervix (Bishop score >5).
2. Decreases the length from the start of the induction until full dilation
3. Decreases the length from the start of the induction until delivery
4. Increases the rate and the speed of spontaneous rupture of membranes (ROM) during cervical ripening
5. Impacts on the rate of cesarean delivery.
6. Impacts on the pain and the satisfaction in women undergoing cervical ripening
7. Impacts on obstetrical and neonatal complications

Study Design:

Prospective, single-center, randomized, two-arm, controlled trial, including women requiring cervical ripening during the process IOL using Balloon catheter

Number of Participants with Rationale:

A total of 290 women will be recruited (145 women in each group) in order to show a reduction in the duration of BC placement, considering a significance criterion set to 0.05 (alpha, two- tailed), and an expected power of at least 90%.

Study procedures:

Patients will be allocated in one of this two groups:

* Intervention or warm group: the BC will be filled with heated saline water up to 40° C
* Standard or room temperature group: the BC will be filled with saline water at room temperature.

In both groups, the insertion of the BC will be done following the same procedure:

The operator will introduce a 14Fr or 18Fr Balloon catheter through the cervical canal, up above the internal orifice using a long Pean clamp and inflate the internal balloon with 30 to 80ml of saline water (NaCl 0.9%) -either heated or unheated, depending on the allocation group- according to the mechanic resistance with a graduated syringe.

Statistical Considerations Main analysis will be performed on an intention-to-treat basis. The main outcome will be evaluated by plotting survival functions according to the allocation group, using the Kaplan-Meier estimator. The associations will be considered as statistically significant when the p-value is below 0.05 (probability of type I error = 0.05). This analysis is also planned for objectives 2 (interval from beginning of IOL and achievement of a favorable cervix) and 3 (interval from beginning of IOL and delivery). For the other outcomes, comparison will be performed using Fisher's exact test, Student's t-test or the Mann-Whitney U test, according to the type of variable.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age at or over 35 weeks
* Singleton pregnancy
* Alive fetus
* Cephalic presentation
* Maternal age ≥ 16 years

Exclusion Criteria:

* Active labor (dilated cervix with spontaneous uterine contractions)
* Prelabor rupture of membranes
* >1 Previous cesarean delivery
* Fetal malformation leading to a possible obstruction of labor (e.g., hydrocephaly, exteriorized fetal tumors, etc.)
* Maternal or fetal disease with indication to accelerate labor (start oxytocin stimulation within 6 hours after insertion of the BC (e.g., pre-eclampsia, chorioamnionitis, etc.)]
* Counterindication to vaginal delivery
* Impossibility to give consent to participation

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
To determine if the use of heated saline in the Balloon Catheter (BC), used for cervical ripening, reduces the length of BC duration, defined as the time from the insertion to spontaneous expulsion or artificial removal of the BC. | Through study completion, an average of 1.5 years
  Duration of BC (i.e., positioning of the transcervical catheter): interval between insertion and retrieval, either after spontaneous expulsion or artificial retrieval.

SECONDARY OUTCOMES:
To evaluate if the use of heated saline compared with room temperature Decreases the length from the start of the induction until the achievement of a favorable cervix (Bishop score >5) | Through study completion, an average of 1.5 years
  Length of cervical ripening phase, defined as the interval between catheter insertion and the achievement of a favorable cervix, defined as Bishop score >5.
Decreases the length from the start of the induction until full dilation | Through study completion, an average of 1.5 years
  Length from the start of the BC insertion until fully dilation
Decreases the length from the start of the induction until the delivery | Through study completion, an average of 1.5 years
  Length from the start of the BC insertion until the delivery
Increases the rate and the speed of spontaneous rupture of membranes (ROM) during cervical ripening | Through study completion, an average of 1.5 years
  Spontaneous rupture of membranes (ROM) during cervical ripening or labor (Yes/No)
  - If Yes, length from the insertion of the BC until spontaneous ROM.
Impacts on the rate of cesarean delivery | Through study completion, an average of 1.5 years
  Mode of delivery (vaginal delivery vs. cesarean delivery)
Impacts on the pain and the satisfaction in women undergoing cervical ripening | Through study completion, an average of 1.5 years
  Pain after catheter insertion assessed using a numeric rating scale (NRS, where NRS = 0 equals no pain and NRS = 10 represents the worst possible pain suffered by the participant). Participants satisfaction of the whole using a five-point Likert scale (1, very dissatisfied; 2, dissatisfied; 3, Enough Satisfied; 4, Satisfied; and 5, very satisfied)
Impacts on obstetrical and neonatal complications | Through study completion, an average of 1.5 years
  Presence of obstetrical complications or neonatal complications

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Genève, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No